CLINICAL TRIAL: NCT01857817
Title: A Randomized, Placebo Controlled, Multicenter Phase 2 Study of Etodolac and Propranolol in Patients With Clinically Progressive Prostate Cancer
Brief Title: Efficacy and Safety Study of Etodolac and Propranolol in Patients With Clinically Progressive Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low patient recruitment
Sponsor: Vicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VT1-SYS-601
Record Dates: First submitted 2013-05-15; First posted 2013-05-20 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Propranolol; Etodolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- VT-122 with physician's choice therapy (Experimental): Participants will receive oral doses of 66 mg propranolol and 680 mg etodolac daily. Propranolol will be administered 44 mg with breakfast and 22 mg in the mid-afternoon (3PM). Etodolac will be administered 340 mg with breakfast and 340 mg with dinner.
  Interventions: Drug: VT-122
- Placebo with physician's choice therapy (Placebo Comparator): Participants will receive physician's choice therapy as the standard of care as well as the placebo capsules that are of the same weight as propranolol and etodolac.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VT-122 — The following will be used in the study for VT-122: propranolol 22 mg immediate-release capsules and etodolac 340 mg capsules.
  Other Names: propranolol; etodolac
  Arms: VT-122 with physician's choice therapy
Drug: Placebo — The placebo capsules will be prepared to match the active drug.
  Arms: Placebo with physician's choice therapy

SUMMARY:
The purpose of this study is to evaluate the clinical benefit of the co-administration of propranolol and etodolac (VT-122 therapy) in patients with clinically progressive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed diagnosis of prostate cancer
2. Male participants who are ≥18 years of age
3. In the opinion of the investigator, the participants have a life expectancy of at least 3 months.
4. Two consecutively rising PSA values or two out of three rising PSA values (2.0 ng/mL is the minimum ending value for PSA) at a minimum of 1-week intervals
5. Have a Karnofsky Performance Score (KPS) equal to or greater than 70
6. Have the following laboratory parameters (may be assessed locally):

   1. Platelet count ≥50 x 10E3/µL
   2. Total bilirubin ≤1.5 mg/dL
   3. Serum creatinine ≤1.5 x upper limit of normal (ULN) or creatinine clearance >60 mL/min calculated using Cockcroft-Gault
   4. Liver enzymes [aspartate transaminase (AST), alanine transaminase (ALT)] ≤2 x ULN
7. Able to provide written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, for any reason without prejudice

Exclusion Criteria:

1. The patient has a history of another primary cancer, with the exception of:

   1. Curatively resected non-melanomatous skin cancer;
   2. Other primary solid tumor with no known active disease presents that in the opinion of the investigator that will not affect patient outcome in the setting of current prostate cancer diagnosis.
2. Contraindication to propranolol, etodolac
3. Patients on beta blockers
4. Patients receiving chemotherapy (e.g., docetaxel, cabazitaxel, taxane, or platinum as single agents or in combination) as their cancer treatment
5. History or evidence of cardiac disease: congestive heart failure; New York Heart Association class 2 or greater; active coronary artery disease; unstable angina, cardiac arrhythmias requiring anti-arrhythmic therapy, atrio-ventricular block of second or third degree, or uncontrolled hypertension, patients with recent (less than 6 months) myocardial infarction (MI) or coronary revascularization
6. Hypotension at the time of screening (i.e., systolic blood pressure less than 110 mmHg. Diastolic blood pressure less than 60 mmHg)
7. Resting heart rate less than 60 bpm at time of screening
8. Any uncontrolled, intercurrent illness that in the opinion of the Investigator may interfere with study evaluation. Participants with uncontrolled diabetes will be excluded from the study.
9. On chronotropic drugs (acetylcholine, digoxin, diltiazem, verapamil, atropine, dopamine, dobutamine, epinephrine, isoproterenol)
10. Active clinically serious infections [> Grade 2 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 4.0]
11. Substance abuse, medical, psychological or social conditions that may, in the opinion of the investigator, interfere with the patient's participation in the study or evaluation of the study results
12. Known or suspected allergy to the investigational agents or any agent given in association with this trial (hypersensitivity reaction, hives, rash, difficulty breathing swelling of your face, lips, tongue, or throat)
13. Any condition that is unstable or which in the opinion of the Investigator could jeopardize the safety of the patient and his/her compliance in the study
14. Patients with uncontrolled diabetes or insulin resistance
15. Participation in any other investigational trial in which receipt of investigational drug or device occurred within 30 days prior to screening for this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in prostate specific antigen (PSA) | baseline (Day 1 Cycle 1) to 12 weeks (Day 1, Cycle 4)

SECONDARY OUTCOMES:
PSA progression | baseline to 12 weeks
PSA doubling time (PSADT) | baseline and every month during treatment
Change in self-reported performance (EQ-5D), pain (visual analog scale [VAS] and opiate usage) | Day 1 Cycle 1, on Day 1 of each subsequent 28-day cycle, and on end of treatment
Time to symptom progression (TTSP) | Day 1 Cycle 1 and Day 1 of each subsequent 28-day cycle
Change in correlative biomarkers | Day 1 Cycle 1, on Day 1 of each subsequent 28-day cycle, and on end of treatment

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Redwood Regional Medical Group, Santa Rosa, California
  - Advanced Urology, Parker, Colorado
  - Manatee Medical Research Institute, LLC, Bradenton, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Midwestern Regional Medical Center, Zion, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Detroit Clinical Research Center, PC, Lansing, Michigan
  - Adult & Pediatric Urology, Sartell, Minnesota
  - AccuMed Research Associates, Garden City, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - Montefiore Medical Center, The Bronx, New York
  - Hendrick Cancer Center, Abilene, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Medical Oncology Associates, PS, Spokane, Washington